CLINICAL TRIAL: NCT06269718
Title: The Changes of Masticatory / Swallowing Functions and Oropharyngeal Muscle Mass on Sonography After Comprehensive Swallowing Training and Tongue - Pressure Resistance Training in Stroke Patients With Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG8N0471
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: stroke; dysphagia; tongue exercises; swallowing therapy; sonography
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The IOPI group (Experimental): tongue muscle strengthening and endurance exercises by using 15-min IOPI biofeedback program. The biofeedback will be 50%-60% of maximal strength
  Interventions: Other: swallowing therapy; Other: IOPI therapy
- The general swallowing group (Active Comparator): oral exercises, tongue movement, and compensatory techniques, swallowing maneuvers and food modifications, will be performed by an experienced speech and language therapist during intervention
  Interventions: Other: swallowing therapy

INTERVENTIONS:
Other: swallowing therapy — oral exercises, tongue movement, and compensatory techniques, swallowing maneuvers and food modifications, will be performed by an experienced speech and language therapist during intervention
Other: IOPI therapy — tongue muscle strengthening and endurance exercises by using 15-min IOPI biofeedback program. The biofeedback will be 50%-60% of maximal strength. (total 1 hour/session for 10 sessions)
  Arms: The IOPI group

SUMMARY:
The aims of this study are:

1. Comparing the ultrasound imaging performance of swallowing and chewing function, tongue pressure and oropharyngeal muscle thickness in stroke patients with different levels of swallowing function
2. To explore the changes in clinical mastication and swallowing functions, tongue pressure and oropharyngeal muscle thickness in patients with dysphagia and stroke after swallowing treatment and neuromuscular electrical stimulation training.
3. To explore the correlation between clinical mastication and swallowing functions, tongue pressure, oropharyngeal muscle thickness and ultrasound imaging results in patients with dysphagia and stroke.

DETAILED DESCRIPTION:
After acute stroke, 25∼45% of patients show difficulties in swallowing, which is associated with a high risk of pneumonia, malnutrition, and mortality. In addition to traditional swallowing therapies for post-stroke dysphagia (PSD), the Iowa Oral Performance Instrument (IOPI) is used to provide tongue exercise program which improving swallowing function. In rehabilitation unit, ultrasound is a convenient tool and is more widely used in investigating oropharyngeal muscles mass and quality in PSD. Therefore, the investigators hope to assess the effects on swallowing function and oropharyngeal muscle mass on sonography after IOPI swallowing training in PSD. In this study, 60 stroke patients with or without dysphagia will be enrolled. Each patient will receive clinical assessments of swallowing and tongue functions, general and oropharyngeal muscles mass and quality by sonography, and life quality. Furthermore, the investigators'll enrolled 50 stroke patients with dysphagia and they will be randomly allocated in two groups. the investigators will provide two interventions including general swallowing therapy, and combined simple and IOPI therapies. First, the investigators will investigate the differences of swallowing and tongue functions, oropharyngeal muscles on sonography in patients with or without PSD. The effects of the swallowing therapies in masticatory and swallowing function, tongue pressure, oropharyngeal muscle mass, and life quality will be explored in PSD by using different swallowing therapies. The investigators will find out the most effective swallowing therapy from these 2 interventions for PSD. Furthermore, the investigators could explore that sonography is a clinically practical tool for assessing oropharyngeal muscles mass and quality in PSD.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients with hemiplegia that are diagnosed with or without dysphagia (FOIS1-7)
* The duration since the onset of stroke should be within 6 months.
* The ages of participants should be from 18 to 80 years old.

Exclusion Criteria:

* The stroke duration is more than 6 months after stroke
* Aged younger than 18 or older than 80 years old
* Any cognitive deficit that leads to communicative difficulty.
* Any other history of systemic diseases that are associated with swallowing difficulty.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
the change from baseline to time of swallowing muscle strength | baseline (before intervention), right after three-week intervention (time 1), and three-week post intervention (time 2) as follow-up assessments
  the evaluation would be executed by an experienced speech and language therapist. The target muscles include tongue and lip strength and endurance.
the change from baseline to time of Masster thickness | baseline (before intervention), right after three-week intervention (time 1), and three-week post intervention (time 2) as follow-up assessments
  The measurement of masseter thickness would be placed at the most prominent area of the masseter muscle in longitudinal and transverse planes.
  The measurements will be taken during relaxation and maximal jaw clenching (2 conditions). The measurements were performed 3 times, and the mean value would be adapted for further analysis.
the change from baseline to time of tongue muscles thickness | baseline (before intervention), right after three-week intervention (time 1), and three-week post intervention (time 2) as follow-up assessments
  For the tongue muscles, the probe will be placed on the point of the lower chin surface be performed at the maximal cross-section area of the muscles in both longitudinal and transverse planes. The measurements were performed 3 times, and expressed as the mean.

SECONDARY OUTCOMES:
the change from baseline to time of general muscle mass | baseline (before intervention), right after three-week intervention (time 1), and three-week post intervention (time 2) as follow-up assessments
  measure bilateral calf circumferences
Measure the change in grip strength (by Jamar hand dynamometer) | baseline (before intervention), right after three-week intervention (time 1), and three-week post intervention (time 2) as follow-up assessments
  the change from baseline to time of general muscle mass
the change from baseline to time of swallowing functions | baseline (before intervention), right after three-week intervention (time 1), and three-week post intervention (time 2) as follow-up assessments
  Functional Oral Intake Scale (FOIS) score is a simple assessing scale to quickly identify the swallowing functions. The score ranges from 1 to 7.
  The score of this scale is defined as follows:
  1, dependency of tube without oral intake ; 2, dependency of tube with inconsistent oral intake; 3, dependency of tube as a supplement with consistent oral intake; 4, total oral intake of a single consistency; 5, total oral intake with specific preparation for multiple consistency; 6, total oral intake without any specific preparation, but avoid specific liquids or food; 7, total oral intake without any restrictions. Higher scores mean a better outcome.
the change from baseline to time of clinical nutrition status | baseline (before intervention), right after three-week intervention (time 1), and three-week post intervention (time 2) as follow-up assessments
  Mini-nutritional assessment short form (MNA) is a screening form to identify patients who are malnourished or at risk of malnutrition, which allows clinicians to intervene earlier to provide adequate nutritional support, prevent further deterioration, and improve patient outcomes.
the change from baseline to time of swallowing functions 100 ml water test | baseline (before intervention), right after three-week intervention (time 1), and three-week post intervention (time 2) as follow-up assessments
  100 ml water test has been used as a screening tool for patients with stroke who are at risk of aspiration. This test could also be used to monitor the complete swallowing performances
the change from baseline to time of quality of life | baseline (before intervention), right after three-week intervention (time 1), and three-week post intervention (time 2) as follow-up assessments
  A self-reported questionnaire, the Dysphagia Handicap Index, would be used to evaluate the quality of life. Dysphagia Handicap Index is for patients with dysphagia that provide information regarding the success or failure of swallowing therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchi Huang, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- ChangGungMH, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No